CLINICAL TRIAL: NCT02651844
Title: Mifepristone Treatment for Breast Cancer Patients Expressing Levels of Progesterone Receptor Isoform A (PRA) Higher Than Those of Isoform B (PRB): Neoadjuvant Therapy.
Brief Title: Mifepristone for Breast Cancer Patients With Higher Levels of Progesterone Receptor Isoform A Than Isoform B.
Acronym: MIPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Provincial Magdalena V. de Martínez (Other)
Collaborators: National Agency for Scientific and Technological Promotion, Argentina (Other); Instituto de Biología y Medicina Experimental (IBYME-CONICET) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIDC-2012-0084
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Progesterone receptor isoforms; Antiprogestins; Mifepristone; Neoadjuvant; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mifepristone (Experimental): Tablets of Mifepristone 200 mg p.o. once a day during 14 days between biopsy and surgery after confirming inclusion criteria
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — At the time a patient enters the protocol, 14 pills will be given to the personnel responsible of giving the patient the medicine at her home (This was a special requirement from the Argentine Authorities).
  Patients and personnel will sign the form each then she gets the medication and after that the signed form will be kept at the CRF file.
  Other Names: RU-486

SUMMARY:
* Seventy per cent of breast cancers express estrogen (ER) and progesterone receptors (PR) and respond to endocrine treatment.
* Actual therapy targets ER.
* There is enough evidence that progestins participate regulating breast cancer growth.
* Antiprogestins block cell proliferation and increase apoptosis in breast cancer models which express high levels of PRA.
* Antiprogestins have been used to treat breast cancer patients that failed to other treatments; benefits were seen in selected patients.
* Mifepristone (MFP) is currently used for medical abortion and for the treatment of Cushing disease.
* MFP might exert agonistic effects when PRB isoform is activated by cAMP. This makes mandatory the evaluation of the PR isoform ratio in breast cancer patients in which MFP is a therapeutic possibility.

Main Goal To evaluate if therapeutic doses of MFP exert beneficial effects on breast cancers expressing levels of PRA higher than those of PRB, evaluated as an inhibition in proliferation markers and/or an increase in apoptotic markers.

* Eligibility

  * Postmenopausal women (one year after menses stop).
  * Women with tumors showing ratios of PRA/PRB higher than 1.5 and PR higher than 50%.
  * Women without previous treatment.
  * All clinical stages with tumors larger than 1.5 cm.
  * Patients without autoimmune diseases and/or asthma.
* Study design

  * Open Interventional.
  * Twenty women will take MFP (200 mg) p.o. once /day during 14 days. As for preliminary studies, to reach this number the investigators will have to evaluate 80-100 patients.
  * Surgery is performed 14 days after treatment initiation, 24 hs after last dose.
  * PR isoform ratio will be evaluated by western blots (WB) in one core biopsy. Additional cores will be used for diagnosis, immunohistochemistry (IHC) of PR, Ki-67 and other markers.
  * At surgery samples will be frozen for molecular studies and fixed and processed for pathological evaluation.
  * Wilcoxon signed rank test will be used to evaluate differences in biomarker expression between core biopsy and surgical samples of each patient.
  * Blood will be collected before treatment initiation and prior to final surgery.
  * Mammographic and echographic studies will be carried out before and after treatment.

DETAILED DESCRIPTION:
Hypothesis

PR are involved in breast cancer growth. The antiprogestin mifepristone (MFP) exerts antitumor effects in mammary carcinomas with high expression of PRA. The investigators hypothesize that breast cancers with higher levels of PRA than PRB will benefit from an antiprogestin therapy.

Precis

The aim of the study is to select 20 breast cancer patients, with primary tumors expressing PR (50% or higher) and 1.5 fold PRA as compared with PRB, for a neoadjuvant treatment with mifepristone (MFP) during 14 days in between biopsy core and surgery. There are no studies at the present time selecting breast cancer patients according to the prevailing PR isoform expressed. This is extremely important since antiprogestins might have no effect or even stimulate those over-expressing PRB.

Background

Breast cancer remains one of the main causes of death in women. Current endocrine treatments are aimed to target either estrogen receptors (ER) or to inhibit the synthesis of 17-β-estradiol (E2). Emerging evidence obtained from experimental studies, as well as from human epidemiology, point to an important role for progestins in breast cancer growth.

Both PR isoforms are transcribed from the same gene. PRB has 933 amino acids while PRA lacks the first 164 amino acids. They play different roles in vivo as demonstrated using knock out models.

MFP, a progesterone antagonist, may also act as an agonist in the presence of PRB. In this context, MFP-bound PR recruit coactivators rather than corepressors. MFP may also exert antiglucocorticoid effects. As an antiprogestin it has been used for different obstetric indications, such as uterine ripening and intrauterine fetal death, at doses higher than 200 mg/day. As an antiglucocorticoid it has potential use in different psychiatric disorders, including depression and Alzheimer's and recently, the FDA approved its use for the treatment of Cushing disease (300 mg daily).

Antiprogestins in breast cancer treatment

The first clinical trial to evaluate antiprogestin therapy in patients recruited 22 patients for a third-line study. Patients were treated with MFP, 200 mg/day, for 1-3 months. There was an 18% response rate following 3 months of therapy. The long-term tolerance was good. Three other studies were reviewed together with unpublished results from a fifth study . There are no other published clinical results for breast cancer treatment using MFP.

More recently, four clinical trials have been recently launched for the evaluation of antiprogestins. The ClinicalTrials.gov Identifier: NCT01138553, testing MFP in neoadjuvancy was discontinued because of difficulties in recruiting and the NCT00555919, Schering, testing lonaprisan, was stopped due to lack of expected clinical response. Two other studies are under way, NCT01800422 testing telapristone and NCT02052128 onapristone.

Antiprogestins in preclinical studies

Using murine mammary carcinomas expressing different PR isoforms, and experimental human breast cancer models manipulated to express different PR ratios, the investigators have demonstrated that only tumors with levels of PRA higher than those of PRB regress with antiprogestin treatment. Moreover, breast cancer samples with higher levels of PRA than PRB respond ex vivo to MFP treatment.

Study design

Registration: The investigators will recruit patients with mammographic and echographic studies that a) have been diagnosed with breast cancer clinically (to be confirmed in biopsy) and b) surgery has been recommended for the treatment of this cancer. Patients will be interviewed by Dr. Gass, and /or Dr. Liguori, or Dr. Paula Martínez-Vazquez, and consented into the study. The original IC will be kept in the CRF of the patient and a copy in the main study file.

Anonymization and generation of the unique patient identifier: Research samples will be anonymized with an identification code. Only Dr. Gass and Dr. Lanari will have access to the codes.

Biopsies: After having signed the IC and having evaluated that the patient is potentially a candidate for the clinical trial, the patient will be biopsied under echographic guide. Three needle cores will be obtained to a) make the final diagnosis, b) measure PRA/PRB isoform ratio by western blot (WB), c) measure ER and PR by immunohistochemistry (IHC) and store the paraffin block for biomarker staining and, d) perform tumor transcriptome. Biopsy core will be flash frozen at -80 °C for molecular studies and the others fixed in 10% buffered formaldehyde for diagnosis determination and PR IHC following routine hospital guidelines.

Blood: Will be collected the same day of biopsy (40 ml by standard hospital procedures) and stored to make different studies in addition to the routine approach: a) MFP measuring b) purify circulating DNA/ microRNAs/tumor cells. This procedure will be repeated the day of surgery.

Diagnosis: Seventy two hours after biopsy, the diagnosis, the PR WB, and the IHC PR value will be available. If the patient qualifies she is ready for the 14 days treatment. All studies will be recorded in the CRF.

Treatment: Generic tablets of MFP 200 mg p.o once a day during 14 days. MFP will be imported from the international pharmacies of Pharma web Canada. Expiration date is July 2018. All medications are manufactured in FDA approved facilities (help@pharmawebcanada.com). Three cases of 99 units each will be purchased. When a patient enters the protocol, 14 pills will be given to the personnel responsible of giving the patient the medicine at her home (requirement from the Argentine Authorities).The form will be signed by patient, worker and by Dr. Gass and the form kept on the patient CRF.

Clinic Control: One week after treatment initiation, patient will go back to the hospital for a clinic control. Note: Due to the extended period of recruitmment, new mifepristone pills were purchased with expiration date October 2019.

Contraindications:

* MFP hypersensitivity.
* Chronic renal failure.
* Asthma.

Side effects: Severe side effects are not expected. Mild effects may include: nausea, vomits, lethargy at low levels. Patients that quit the protocol will be treated as those inside the protocol.

Contraindicated therapies: If women are taking other medication, the attending physicians will evaluate possible interactions case by case. The patient will be excluded from the protocol if needed. The patients will be instructed to notify the attending physician should the necessity arises to be put under a medication different from that administered as part of the trial.

Before surgery: New mammogram and ecography to compare images before and after treatment (no differences expected).

Surgery: Under routine Hospital guidelines for all breast cancer patients. It will be performed on day 15 after treatment initiation. Tissue will be collected for immunohistochemical staining (formalin fixed) and kept frozen at -80°C for genomic/proteomic studies. Blood will also collected as mentioned before.

Technical Procedures

Sample transport: Anonymized frozen samples will be sent to IBYME for WB studies in dry ice using a special transport Enterprise (Transportes Ambientales S.A). At IBYME Security personnel will record the arrival and then transported to the LCH Lab.

PR WB: Nuclear extracts will be performed and processed as described previously. T47D cells will be used as a positive control. Paola Rojas will be in charge of the determination of the PRA/PRB ratio. Procedures will be recorded. Results will be sent to Dr.Liguori and Dr. Gass, and a copy of them will be kept in the CRF.

PR IHC: Five micron paraffin embedded core tissues will be processed for standard PR IHC assays using FDA approved antibodies and quantified as described previously. Two pathologists (Dr. Gonzalez and Dr. May, supervised by Dr. Molinolo) will quantify and score the IHC staining. The pathologists will inform the PR score to Dr. Liguori, 72 hs after biopsy who will include the record at the patient CRF.

Decision for patient inclusion: Dr Liguori will be responsible of collecting the WB info and the PR IHC info and Dr. Gass will have to agree that the patient might enter the protocol because she matches with all the inclusion criteria. A signed form will be included at the patient CRF.

Biomarker evaluation: All assays for primary and secondary endpoints will be analyzed after concluding with patient recruitment. Nuclear Ki-67 staining will be evaluated according to Goldhirsch et al., 2013, and other biomarkers will be evaluated at the end of the study comparing biopsy and surgery scores of all patients recruited. Cytoplasmic, nuclear and membrane stainings will also be considered for biomarkers other than hormone receptors and Ki-67. Tumors with Ki-67 scoring differences greater than 10% between the two pathologists will be reevaluated until complete agreement is obtained. For differences less than 10%, the average score will be considered. If a positive response is seen (30% change in biomarker expression between biopsy and surgery), the investigators will start with the molecular analysis of the samples using available genomic platforms.

Statistics: Descriptive statistics will be used to summarize subject baseline characteristics, treatment administration/compliance, etc. Data will also be displayed graphically, when appropriate. An accounting of all subjects enrolled will be summarized. The number of subjects discontinuing from the study and the reasons for discontinuation will be tabulated. Subjects who did not meet eligibility criteria will be described. Demographic and baseline characteristics such as subject age, sex, race, height, weight, ECOG performance status, malignancy history, and medical history will be summarized. Wilcoxon signed rank test will be used to compare changes in biomarker expression.

Number of patients to be included: To calculate the number of patients to be included, the investigators fixed Type 1 error: 0.05 and Type 2: 0.10, Power 0.8. It was assumed that no differences should be registered between biopsy and surgery in the Ki-67 or apoptotic indices in the absence of treatment and considered a 30% decrease in Ki-67 a positive result. Unpublished data suggest that 37.3% of patients have PRA/PRB higher than 1.5 indicating that around 80 biopsies will be studied by WB to meet the right number.

Insurance: Prudencia Seguros, # 00056924 hired by the Hospital

Documents to include in the regulatory File:

1. Argentina Health Ministry Regulation Res 1480 ANMAT
2. Last version of the protocol presented to the ANMAT (version 3; March 16 2015)
3. Versions approved by clinicaltrials.gov
4. Model of IC
5. Participants CV
6. IRBs approvals and amendments
7. ANMAT form accepting drug importation
8. All forms related to medication administration mentioned previously
9. Documents related to the certification of the IRBs
10. Protocols concerning WB and IHC including methods of equipment calibration
11. SOP related to all clinical practice

The entire file will be available for possible inspection by the Institutional IRB or MINCYT, CONICET or other authorities who may be concerned. Dr. Gass will be responsible for providing all the data requested by the evaluating committees.

Notes: Dr M. Liguori is no longer in charge of the patients since August 2018. Dr Hugo Gass is in charge of patient recruitment, biopsies and clinic evaluation. Dr. Marìa May and Dr. Pedro Gonzalez, pathologists, are no longer involved in the study. They were replaced by Eunice Spengler and Silvia Ines Vanzulli.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  1. Postmenopausal women (one year after menses stop)
  2. Confirmed diagnosis of breast cancer
  3. Tumors with higher expression PR > 50 % measured by IHC and PRA/RPB ratio equal or higher than 1.5 measured by WB
  4. All clinical stages with tumor size greater than 1.5 cm to allow obtaining material from biopsy cores
  5. OMS condition: 1 Adequate function of organs and systems

Hematopoietic parameters:

* Hemoglobin: 10 gr/mL
* Neutrophil counting: 1.500/mm3
* CD4 counting: 400/mm3
* Platelets counting: 100.000/mm3 Liver parameters
* Total albumin: 1.5 fold normal limit
* AST/ALT: 1.5 fold normal limit Renal
* Creatinine: 1.5 fold normal limit 6. Absence of other controlled disease 7. Patients willing to sign consent

Exclusion Criteria:

* Exclusion criteria

  1. Patients with no recommended surgery
  2. Patients which have received any other treatment for this cancer
  3. Patients expressing ER but expressing PRA/PRB levels lower than 1.5
  4. Hepatitis infection (HBV o HCV)
  5. HIV infection.
  6. Cognitive alterations which limit the understanding of the protocol or compliance to the protocol
  7. Prolonged QT/QTc basal interval

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Measurable decrease in tumor cell proliferation from baseline to time of surgery | Baseline to time of surgery (14 days of treatment between biopsy core and surgery)
  Treatment efficacy will be assessed by comparing tissue samples from the baseline biopsy and tissue samples collected from the day of surgery, evaluating if there is a decrease in the proliferating index (Ki-67 expression by immunohistochemistry). Positive response: differences higher than 30%.

SECONDARY OUTCOMES:
Measurable increases in apoptotic markers from baseline to time of surgery | Baseline to time of surgery (14 days of treatment between biopsy core and surgery)
  Treatment efficacy will be assessed by comparing tissue samples from the baseline biopsy and tissue samples collected from the day of surgery, evaluating if there is an increase in apoptotic cells measuring TUNNEL and caspase 3 expression. Positive response: difference higher than 30%.
Measurable changes in signaling pathways downstream PR | Baseline to time of surgery (14 days of treatment between biopsy core and surgery)
  MFP action will be measured evaluating the expression of downstream markers related to PR activation such as CCND1, MYC, pSTAT5 and other proteins by immunohistochemistry. Positive response: differences higher than 30%

OTHER OUTCOMES:
Changes in tumor size | Baseline to time of surgery (14 days of treatment between biopsy core and surgery)
  Measured by ecographic imaging. Twenty per cent of decrease in overall tumor size will be considered as a significant change.
RNAseq analysis of gene expression and Proteomics to evaluate possible deregulated pathways | Baseline to time of surgery (14 days of treatment between biopsy core and surgery)
  Differences in gene and protein expression between biopsy core and surgery sample higher than 20 % will be considered as an effective drug response.
Measure serum Mifepristone levels after 7/14 days Mifepristone treatment and other steroid hormone precursors | Baseline to time of surgery (14 days of treatment between biopsy core and surgery), and an intermediate timepoint
  Levels of Mifepristone and other steroids will be measured by HPLC or LC-MS/MS in the blood sample after treatment and correlate these levels with response to treatment (outcome 1).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lanari, PhD, Study Director — IBYME-CONICET
Locations (1):
- HospitalPMVM, General Pacheco, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lanari C, Wargon V, Rojas P, Molinolo AA. Antiprogestins in breast cancer treatment: are we ready? Endocr Relat Cancer. 2012 May 3;19(3):R35-50. doi: 10.1530/ERC-11-0378. Print 2012 Jun. PMID 22351709
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Hofseth LJ, Raafat AM, Osuch JR, Pathak DR, Slomski CA, Haslam SZ. Hormone replacement therapy with estrogen or estrogen plus medroxyprogesterone acetate is associated with increased epithelial proliferation in the normal postmenopausal breast. J Clin Endocrinol Metab. 1999 Dec;84(12):4559-65. doi: 10.1210/jcem.84.12.6194. PMID 10599719
- [Background] Greiser CM, Greiser EM, Doren M. Menopausal hormone therapy and risk of breast cancer: a meta-analysis of epidemiological studies and randomized controlled trials. Hum Reprod Update. 2005 Nov-Dec;11(6):561-73. doi: 10.1093/humupd/dmi031. Epub 2005 Sep 8. PMID 16150812
- [Background] Chlebowski RT, Hendrix SL, Langer RD, Stefanick ML, Gass M, Lane D, Rodabough RJ, Gilligan MA, Cyr MG, Thomson CA, Khandekar J, Petrovitch H, McTiernan A; WHI Investigators. Influence of estrogen plus progestin on breast cancer and mammography in healthy postmenopausal women: the Women's Health Initiative Randomized Trial. JAMA. 2003 Jun 25;289(24):3243-53. doi: 10.1001/jama.289.24.3243. PMID 12824205
- [Background] Beral V; Million Women Study Collaborators. Breast cancer and hormone-replacement therapy in the Million Women Study. Lancet. 2003 Aug 9;362(9382):419-27. doi: 10.1016/s0140-6736(03)14065-2. PMID 12927427
- [Background] Kastner P, Krust A, Turcotte B, Stropp U, Tora L, Gronemeyer H, Chambon P. Two distinct estrogen-regulated promoters generate transcripts encoding the two functionally different human progesterone receptor forms A and B. EMBO J. 1990 May;9(5):1603-14. doi: 10.1002/j.1460-2075.1990.tb08280.x. PMID 2328727
- [Background] Lydon JP, Ge G, Kittrell FS, Medina D, O'Malley BW. Murine mammary gland carcinogenesis is critically dependent on progesterone receptor function. Cancer Res. 1999 Sep 1;59(17):4276-84. PMID 10485472
- [Background] Jackson TA, Richer JK, Bain DL, Takimoto GS, Tung L, Horwitz KB. The partial agonist activity of antagonist-occupied steroid receptors is controlled by a novel hinge domain-binding coactivator L7/SPA and the corepressors N-CoR or SMRT. Mol Endocrinol. 1997 Jun;11(6):693-705. doi: 10.1210/mend.11.6.0004. PMID 9171233
- [Background] Wargon V, Riggio M, Giulianelli S, Sequeira GR, Rojas P, May M, Polo ML, Gorostiaga MA, Jacobsen B, Molinolo A, Novaro V, Lanari C. Progestin and antiprogestin responsiveness in breast cancer is driven by the PRA/PRB ratio via AIB1 or SMRT recruitment to the CCND1 and MYC promoters. Int J Cancer. 2015 Jun 1;136(11):2680-92. doi: 10.1002/ijc.29304. Epub 2014 Nov 12. PMID 25363551
- [Background] Ulmann A, Dubois C. Anti-progesterones in obstetrics, ectopic pregnancies and gynaecological malignancy. Baillieres Clin Obstet Gynaecol. 1988 Sep;2(3):631-8. doi: 10.1016/s0950-3552(88)80049-x. PMID 3069266
- [Background] Benagiano G, Bastianelli C, Farris M. Selective progesterone receptor modulators 3: use in oncology, endocrinology and psychiatry. Expert Opin Pharmacother. 2008 Oct;9(14):2487-96. doi: 10.1517/14656566.9.14.2487. PMID 18778186
- [Background] Fleseriu M, Biller BM, Findling JW, Molitch ME, Schteingart DE, Gross C; SEISMIC Study Investigators. Mifepristone, a glucocorticoid receptor antagonist, produces clinical and metabolic benefits in patients with Cushing's syndrome. J Clin Endocrinol Metab. 2012 Jun;97(6):2039-49. doi: 10.1210/jc.2011-3350. Epub 2012 Mar 30. PMID 22466348
- [Background] Romieu G, Maudelonde T, Ulmann A, Pujol H, Grenier J, Cavalie G, Khalaf S, Rochefort H. The antiprogestin RU486 in advanced breast cancer: preliminary clinical trial. Bull Cancer. 1987;74(4):455-61. PMID 3311238
- [Background] Klijn JG, Setyono-Han B, Foekens JA. Progesterone antagonists and progesterone receptor modulators in the treatment of breast cancer. Steroids. 2000 Oct-Nov;65(10-11):825-30. doi: 10.1016/s0039-128x(00)00195-1. PMID 11108894
- [Background] Jonat W, Bachelot T, Ruhstaller T, Kuss I, Reimann U, Robertson JFR. Randomized phase II study of lonaprisan as second-line therapy for progesterone receptor-positive breast cancer. Ann Oncol. 2013 Oct;24(10):2543-2548. doi: 10.1093/annonc/mdt216. Epub 2013 Jun 20. PMID 23788750
- [Background] Wargon V, Helguero LA, Bolado J, Rojas P, Novaro V, Molinolo A, Lanari C. Reversal of antiprogestin resistance and progesterone receptor isoform ratio in acquired resistant mammary carcinomas. Breast Cancer Res Treat. 2009 Aug;116(3):449-60. doi: 10.1007/s10549-008-0150-y. Epub 2008 Aug 3. PMID 18677559
- [Background] Wargon V, Fernandez SV, Goin M, Giulianelli S, Russo J, Lanari C. Hypermethylation of the progesterone receptor A in constitutive antiprogestin-resistant mouse mammary carcinomas. Breast Cancer Res Treat. 2011 Apr;126(2):319-32. doi: 10.1007/s10549-010-0908-x. Epub 2010 May 4. PMID 20440553
- [Background] Vanzulli S, Efeyan A, Benavides F, Helguero LA, Peters G, Shen J, Conti CJ, Lanari C, Molinolo A. p21, p27 and p53 in estrogen and antiprogestin-induced tumor regression of experimental mouse mammary ductal carcinomas. Carcinogenesis. 2002 May;23(5):749-58. doi: 10.1093/carcin/23.5.749. PMID 12016147
- [Background] Hammond ME, Hayes DF, Dowsett M, Allred DC, Hagerty KL, Badve S, Fitzgibbons PL, Francis G, Goldstein NS, Hayes M, Hicks DG, Lester S, Love R, Mangu PB, McShane L, Miller K, Osborne CK, Paik S, Perlmutter J, Rhodes A, Sasano H, Schwartz JN, Sweep FC, Taube S, Torlakovic EE, Valenstein P, Viale G, Visscher D, Wheeler T, Williams RB, Wittliff JL, Wolff AC. American Society of Clinical Oncology/College Of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer. J Clin Oncol. 2010 Jun 1;28(16):2784-95. doi: 10.1200/JCO.2009.25.6529. Epub 2010 Apr 19. PMID 20404251
- [Background] Goldhirsch A, Winer EP, Coates AS, Gelber RD, Piccart-Gebhart M, Thurlimann B, Senn HJ; Panel members. Personalizing the treatment of women with early breast cancer: highlights of the St Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2013. Ann Oncol. 2013 Sep;24(9):2206-23. doi: 10.1093/annonc/mdt303. Epub 2013 Aug 4. PMID 23917950
- [Derived] Elia A, Saldain L, Lovisi S, Martinez Vazquez P, Burruchaga J, Lamb CA, Luthy IA, Diez F, Homer NZM, Andrew R, Rojas P, Lanari C. Steroid profile in patients with breast cancer and in mice treated with mifepristone. Endocr Relat Cancer. 2023 Dec 13;31(2):e230238. doi: 10.1530/ERC-23-0238. Print 2024 Feb 1. PMID 37962553
- [Derived] Elia A, Saldain L, Vanzulli SI, Helguero LA, Lamb CA, Fabris V, Pataccini G, Martinez-Vazquez P, Burruchaga J, Caillet-Bois I, Spengler E, Acosta Haab G, Liguori M, Castets A, Lovisi S, Abascal MF, Novaro V, Sanchez J, Munoz J, Belizan JM, Abba MC, Gass H, Rojas P, Lanari C. Beneficial Effects of Mifepristone Treatment in Patients with Breast Cancer Selected by the Progesterone Receptor Isoform Ratio: Results from the MIPRA Trial. Clin Cancer Res. 2023 Mar 1;29(5):866-877. doi: 10.1158/1078-0432.CCR-22-2060. PMID 36269797